CLINICAL TRIAL: NCT00216723
Title: Efficacy and Safety of Aripiprazole in Patients With Schizophrenia or Bipolar Disorder
Status: Completed | Type: Observational
Sponsor: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Seo Bo Yeon, Korea Otsuka Pharmaceutical Co.,Ltd.
Other Study IDs: Korea Abilify PMS
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2013-10-23 (Estimated); Status verified 2013-10

CONDITIONS: Schizophrenia; Bipolar Disorder
Keywords: Aripiprazole; Schizophrenia; Bipolar Disorder
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder | interventions — Aripiprazole

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective

INTERVENTIONS:
Drug: Aripiprazole — The recommended starting and target dose for Abilify is 10 or 15mg/day administered on a once-a-day schedule without regard to meals.
  (Administer 10 to 30 mg/day according to the patient's condition)

SUMMARY:
This is a multicenter,open-label,prospective study of Aripiprazole use in patients with schizophrenia and bipolar disorder.

DETAILED DESCRIPTION:
This is a multicenter,open-label,prospective study of Aripiprazole use in patients with schizophrenia and bipolar disorder.

Qualified schizophrenia patients will be enrolled to an 12-week treatment phase of Aripiprazole by physician's assessment.

Qualified bipolar disorder patients will be enrolled to an 8-week treatment phase of Aripiprazole by physician's assessment.

This study will be continued for 6 years. The final report of Aripiprazole PMS will be submitted to KFDA on December 28, 2009.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a schizophrenia or schizoaffective disorder or bipolar disorder according to DSM-IV criteria
* Age: more than 18 years of age

Exclusion Criteria:

* Unqualified patients judged by study investigator(s)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patient with a schizophrenia or schizoaffective disorder or bipolar disorder according to DSM-IV criteria
  * Age: more than 18 years of age
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2004-04; Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jieun Kwon, Study Director — Korea Otsuka Pharmaceutical Co., Ltd.
Locations (2):
- South Korea (2):
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul